



**NHS Foundation Trust** 

**Royal Free Hospital** 

3<sup>rd</sup> Floor Renal Research Office Pond Street

London NW32QG

Tel: 020 7472 6687

## Study ID: Recipient \_ \_ \_ Donor \_ \_ \_

## **CONSENT FORM**

## Longitudinal characterisation of the host microbiota after kidney donation and transplantation

| Chief I | nvestigator: Mr Reza Motallebzade | h | ., | |
|---|---|---|---|---|
| | _ | | | Please initial each box |
| 1. | during the study may be looked at by responsible individuals from Royal Free London NHS Foundation Trust or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | 2 | |
| | | | • | ed on on one on one on one one one one one |
| | | | Royal Free London evant to my taking | |
| 4. | | | • • | |
| 5. | <ol> <li>I agree to my samples being used as described in the information sheet and I understand that the anonymised samples may be processed and analysed at laboratories of named collaborators outside Royal Free Hospital &amp; UCL as justified by the expertise and resources required to meet the objectives of this study.</li> <li>I agree to my samples being used for future ethically approved non-commercial research studies related to the clinical condition(s) of this study</li> <li>I agree to my blood and biopsy samples being used for genetic (RNA/DNA) analysis [optional]</li> </ol> | | | t<br>, |
| 6. | | | | |
| 7. | | | | |
| 8. | . I understand that the anonymised results from the study will be published in peer review journals and will be presented both nationally and internationally. | | | |
| 9. | I agree to take part in the above st | udy. | | |
| Name of Patient | | <br>Date | Signature | 2 |
| | | | Signature | |
| Name of person taking consent | | Date | Signatiire | د |

When completed, 1 original for patient; 1 for the site file; 1 (original) to be kept with hospital notes (i.e. scanned into EDRM at RFL)

